CLINICAL TRIAL: NCT03244631
Title: Prospective, Single Blind Randomzied Controlled Trial Comparing Lumbar Plexus Peripheral Nerve Block Versus Peri-capsular Injection for Hip Arthroscopy
Brief Title: Pain Control in Hip Arthroscopy: Comparing Lumbar Plexus Versus Peri-capsular Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington Orthopaedics and Sports Medicine (Other)
Responsible Party: Principal Investigator, Andrew B. Wolff, MD, Attending Surgeon, Washington Orthopaedics and Sports Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20171307
Record Dates: First submitted 2017-07-28; First posted 2017-08-09 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Nerve Block; Hip Arthroscopy

STUDY DESIGN:
Intervention Model Description: Prospective randomized
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumbar Plexus Block (Active Comparator): A lumbar plexus 'nerve block' is a procedure in which local anesthetic ("numbing medicine") is injected around a specific group of nerves to provide pain relief directly to the nerves supplying the area of the body undergoing surgery.
  Interventions: Procedure: Lumbar Plexus BLock
- Pericapsular Injection (Active Comparator): The pericapsular injection is a procedure in which local anesthetic ("numbing medicine") is injected around the hip joint to provide direct pain relief to the area undergoing surgery.
  Interventions: Procedure: Pericapsular injection

INTERVENTIONS:
Procedure: Lumbar Plexus BLock — Peripheral nerve block
  Arms: Lumbar Plexus Block
Procedure: Pericapsular injection — Injection around the area undergoing surgery
  Arms: Pericapsular Injection

SUMMARY:
Comparison of lumbar plexus nerve block versus pericapsular injection for pain control during hip arthroscopy

DETAILED DESCRIPTION:
The purpose of this study is to compare two different methods of pain control during and after hip arthroscopy surgery. It is not clear which of many different pain control methods are ideal to reduce pain for patients; consequently, the investigators are performing this study to compare the two main choices for pain control commonly used in order to identify if either is superior to the other.

ELIGIBILITY:
Inclusion Criteria:

1. Patient scheduled to undergo hip arthroscopy with Dr. Wolff
2. Patient age between 25 and 60 years of age.

Exclusion Criteria:

1. Patient has known allergy to ropivicaine or morphine.
2. Patient unable to speak/read English (No translators available in clinic site).
3. Pregnant female.
4. Patient has a pre-operative narcotic use for hip pain
5. Patient has pre-existing chronic pain disorder (i.e. fibromyalgia)

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Pain score | At the one hour point in the PACU
  Compare post-operative pain scores in the immediate post-operative period as defined by visual-analog pain scale at the time point of one hour spent in the post-anesthesia care unit (PACU).

SECONDARY OUTCOMES:
Morphine equivalents | At the two hour point in the PACU
  Compare the total morphine equivalents of opioids provided in the PACU within the first two hours of time spent in the PACU
Time spent in PACU | Immediately after surgery
  Compare the overall time spent in the PACU as defined by time to arrival to time to discharge vitals.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wolff, MD, Principal Investigator — Washington Orthopaedics and Sports Medicine
Locations (1):
- Washington Orthopedics and Sports Medicine, Chevy Chase, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scanaliato JP, Christensen D, Polmear MM, Salfiti C, Gaspar PS, Wolff AB. Prospective Single-Blinded Randomized Controlled Trial Comparing Pericapsular Injection Versus Lumbar Plexus Peripheral Nerve Block for Hip Arthroscopy. Am J Sports Med. 2020 Sep;48(11):2740-2746. doi: 10.1177/0363546520943580. Epub 2020 Aug 6. PMID 32757999